CLINICAL TRIAL: NCT02833246
Title: Using a Patient-Centered mHealth Intervention to Improve Adherence to Oral Anticancer Medications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16-810
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Sarcoma; Lung; Solid Tumor Gastrointestinal
Keywords: texting; Adherence to Oral Anticancer Medications; 16-810
MeSH Terms: conditions — Sarcoma

ARMS (2):
- SMS/MMS text messaging (Experimental): Patients will be able to tailor their SMS/MMS reminders with respect to when (i.e., what time of day) they wish to receive the reminders, as well as how often the messages are sent (e.g., morning and evening).
  Interventions: Other: SMS/MMS text messaging
- usual care (Active Comparator): This includes physician and nursing assessment and intervention for any identified AEs. Of note, there is not currently standard follow-up that patients receive from nursing or physician staff while on an OAM treatment. Patients are encouraged to call their physician's office with any questions or changes in their medical status but are not called routinely by MSK staff.
  Interventions: Other: usual care

INTERVENTIONS:
Other: SMS/MMS text messaging — text messaging reminders on oral chemotherapy medication adherence
  Arms: SMS/MMS text messaging
Other: usual care
  Arms: usual care

SUMMARY:
This study is being done to determine if sending reminder text messages helps patients take their Oral Anticancer Medication (OAMs) when they are supposed to.

ELIGIBILITY:
Inclusion Criteria:

* Patient in the Sarcoma, Solid Tumor Gastrointestinal (ST GI), and Thoracic Medicine service at MSK.
* Starting a new treatment regimen that includes a single oral anticancer medication
* Patients must have a mobile phone that can send and receive SMS/MMS messages and is internet-enabled.
* Age 18 or older.
* Ability to speak and read English because we do not have the resources to translate the text messages into other languages.

Exclusion Criteria:

* Patient expresses inability or unfamiliarity with using SMS/MMS messaging on their phone and is unwilling to be trained in the use of this technology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-06-28 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2018-11-14 (Actual)

PRIMARY OUTCOMES:
objective pill count | 1 year
  is greater or less than the amount of OAM that the patient should have in their possession.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Atkinson, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/